CLINICAL TRIAL: NCT07260331
Title: The Role of Musical Stimulation Intensity on Postural Control in Athletes: A Virtual Reality-Based Posturography Study
Brief Title: Musical Stimulation Intensity and Postural Control (MUSIC-POST)
Acronym: MUSIC-POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanifi Korkmaz (Other)
Responsible Party: Sponsor-Investigator, Hanifi Korkmaz, Asst. Prof. Dr., Malatya Turgut Ozal University
Organization: Malatya Turgut Ozal University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2025/95; 2025/95 (Other: MTÜ Health Sciences Ethics Committee)
Record Dates: First submitted 2025-11-15; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Health Adult Subjects; Adults; Athlete
Keywords: Postural Stability; Virtual Reality; Auditory Intensity

STUDY DESIGN:
Intervention Model Description: This is a single-arm crossover design where all participants sequentially complete balance tests under three auditory intensity conditions (low, medium, high). Randomization refers only to the order of condition presentation.
Masking Description: Although the study includes three auditory intensity conditions (low, medium, high), all participants are enrolled in a single group undergoing a crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auditory Stimulation Conditions (Experimental): Participants completed balance assessments under three auditory intensity conditions: low (40 dB), medium (70 dB), and high (90 dB). Each condition was administered in a randomized crossover design using a virtual reality-based (VR) posturography system. Washout periods were included to prevent carryover effects.
  Interventions: Device: Virtual Reality-Based Auditory Stimulation

INTERVENTIONS:
Device: Virtual Reality-Based Auditory Stimulation — Participants performed postural control tasks using a virtual reality-based posturography system under three auditory intensity conditions (low, medium, high). Controlled auditory stimuli were delivered via headphones, and balance performance was recorded for each condition.
  Other Names: BalanceVR Posturography

SUMMARY:
This study aims to investigate the effects of musical stimulation intensity on postural control in athletes using a virtual reality-based (VR) static posturography system. Athletes from various sports disciplines will be exposed to low-, medium-, and high-intensity music during balance assessments. The study will analyze changes in postural stability parameters under different auditory stimulation levels to understand the interaction between auditory processing, proprioception, and motor control in athletes.

DETAILED DESCRIPTION:
This experimental study aims to examine the role of musical stimulation intensity on postural control performance in athletes through a virtual reality (VR)-based static posturography system. The study will include athletes from different sports disciplines such as volleyball, football, swimming, tennis, and combat sports.

Participants will perform balance tests under three controlled auditory conditions: low-, medium-, and high-intensity music. The VR-based posturography device will provide immersive visual feedback and precise measurements of Center-of-Pressure (COP) displacement, reaction time, and directional control. The auditory stimuli will be delivered through headphones integrated into the VR headset to ensure standardized sound intensity levels.

The primary outcome measures include changes in stability indices, sensory organization, and Limits of Stability (LOS) parameters across the three music intensity conditions. Secondary outcomes will analyze the relationship between noise sensitivity scores and postural control metrics.

This study will contribute to understanding how auditory stimulation interacts with sensorimotor integration and balance control mechanisms in athletes. The findings may support the design of VR-based training and rehabilitation programs that integrate controlled auditory environments to optimize performance and postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years

Actively training in sports (minimum 3 sessions per week)

Normal hearing thresholds (≤20 dB HL at 0.5-8 kHz)

No history of vestibular, neurological, or musculoskeletal disorders

Voluntary participation and informed consent

Exclusion Criteria:

* Any diagnosed balance or vestibular disorder

History of ear surgery or chronic otitis media

Current use of medications affecting balance or cognition

Exposure to intense noise or ototoxic substances in the past month

Refusal to participate or inability to complete VR-based testing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Postural Stability Score measured by VR-based Static Posturography | Assessed after each condition within one testing session (~30 minutes).
  Postural Stability Score (%) obtained from VR-based static posturography during balance tasks under low, medium, and high auditory intensity conditions. The score reflects overall postural steadiness based on center-of-pressure displacement metrics.

SECONDARY OUTCOMES:
Mean Velocity measured by VR-based Posturography | Recorded immediately after each test condition within a single session (≈35 minutes per participant).
  Mean velocity of center-of-pressure sway was recorded using a VR-based static posturography system under low (40 dB), medium (70 dB), and high (90 dB) auditory intensity conditions to examine auditory effects on dynamic postural adjustments.
Reaction Time measured by VR-based Static Posturography | Recorded immediately after each test condition within a single session (≈35 minutes per participant).
  Motor reaction time to initiate movement toward visual targets was recorded using a VR-based static posturography system under low (40 dB), medium (70 dB), and high (90 dB) auditory intensity conditions to determine the influence of auditory intensity on movement initiation.
Endpoint Excursion measured by VR-based Static Posturography | Recorded immediately after each test condition within a single session (≈35 minutes per participant).
  Maximum endpoint excursion toward visual targets was recorded using a VR-based static posturography system under low (40 dB), medium (70 dB), and high (90 dB) auditory intensity conditions to evaluate how musical stimulation intensity affected the accuracy of voluntary postural movements.
Directional Control measured by VR-based Static Posturography | Recorded immediately after each test condition within a single session (≈35 minutes per participant).
  Directional control values reflecting movement efficiency toward visual targets were recorded using a VR-based static posturography system under low (40 dB), medium (70 dB), and high (90 dB) auditory intensity conditions to examine whether sound intensity influenced movement accuracy and postural strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Hanifi Korkmaz, pHD, Principal Investigator — Malatya Turgut Özal University, Vocational School of Health Services, Department of Child Care and Youth Services
Locations (1):
- Malatya Training and Research Hospital, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy regulations and institutional data protection policies. The dataset includes sensitive personal information collected under specific ethical approval limited to the research team.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT07260331/Prot_SAP_000.pdf